CLINICAL TRIAL: NCT03631537
Title: Effect of Nutrition-support-team Based Intervention on Nutritional Status, Chemotherapy Tolerance and Prognosis in Patients With Advanced Gastrointestinal Cancer
Brief Title: Nutrition-support-team Based Intervention in Patients With Advanced Gastrointestinal Cancer
Acronym: NSTBIPAGC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJTU1AF-CRF-2017-027
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2017-11

CONDITIONS: Malnutrition; Gastrointestinal Cancer; Nutrition Aspect of Cancer
MeSH Terms: conditions — Malnutrition; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Study group: receive nutritional intervention from the nutritional support team; Control group: receive routine nutritional support from clinicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NST group (Experimental): Nutrition support team gives the dietary supplement or other nutritional support during the period of chemotherapy
  Interventions: Other: NST group
- routine group (No Intervention): clinicians decide whether to give and how to give the dietary supplement and other nutritional support

INTERVENTIONS:
Other: NST group — Nutrition-support-team based intervention on nutrition, including dietary supplement, parenteral nutrient solutions and patient education
  Arms: NST group

SUMMARY:
The research studies patients with advanced gastrointestinal cancer who receive chemotherapy in the medical oncology department of the First Affiliated Hospital of Xian Jiaotong University. All patients receive the nutritional risk assessment by the nutritional support team first, and patients with nutritional risk or malnutrition are randomly assigned to the study group and the control group. The study group receive nutritional intervention from the nutritional support team during the period of chemotherapy, while the control group receive routine nutritional support from their clinicians. In the control group, nurses execute the doctors' advice on nutrition, and the nutrition support team does not actively communicate with doctors about the nutritional risk of patients or interfere with it. The baseline characteristics, chemotherapy efficacy, adverse events and prognosis are collected in both groups. At last, data are analyzed to clarify the nutritional status and related factors of patients with advanced gastrointestinal cancer in our hospital, and most important to explore the effect of nutrition-support-team intervention on nutritional status, chemotherapy tolerance and prognosis of patients with advanced gastrointestinal cancer.

DETAILED DESCRIPTION:
Baseline data include age, gender, pain, sleep condition, family care, tumor type, tumor stage, combined disease, chemotherapy regimen and concomitant medication.

Nutritional risk assessments are performed by the nutrition support team just after enrollment, every two cycles of chemotherapy and at the end of the study. The adverse events of chemotherapy are collected and recorded at the end of each cycle. CT or MRI is performed to evaluate efficacy of chemotherapy every two treatment cycles. Patient after one treatment cycle can receive CT or MRI in advance if the clinical condition is worsening.

ELIGIBILITY:
Inclusion Criteria:

* advanced (recurrent or metastatic) gastrointestinal malignancies confirmed by pathology, plan to be treated with chemotherapy
* the expected life period is more than 3 months
* did not receive chemotherapy, radiotherapy, molecular targeted therapy or surgery in the last 4 weeks
* has been recovered from the acute toxicity of previous treatment (if patient received surgery, the wound must have completely healed)
* at least one measurable lesion according to RECIST 1.1 edition (the measurable lesion has not received radiotherapy)
* normal function of main organs:Blood routine examination needs to be met: Hb≥90g/L (without blood transfusions within 14 days); ANC≥1.5×109/L; PLT≥80×109/LBiochemical examination should conform to the following standards: TBIL≤1.5×ULN (upper limit of normal value); ALT and AST≤2.5×ULN (ALT and AST≤5×ULN, in case of liver metastasis); Serum creatinine ≤1×ULN, creatinine clearance rate >50ml/min (Cockcroft-Gault formula)
* volunteer to participate in the study, sign the informed consent, and cooperate with good compliance

Exclusion Criteria:

* pregnancy or lactation
* having a long-term unhealed wound, traumatic or pathological fracture
* urinary protein > 2+ or 24 hour urinary protein >1.0g
* suffering from mental illness
* with hypertension and fail to get good control through antihypertensive medication (systolic pressure >140mmHg and/or diastolic pressure >90mmHg)
* serious diabetes, heart disease (including but not limited to myocardial ischemia, myocardial infarction, cardiac insufficiency, congestive heart failure), thrombotic diseases (including but not limited to cerebral hemorrhage, deep venous thrombosis and pulmonary embolism)
* long-term use of steroid for other medical reasons
* with diseases that may increasing the underlying research risk judged by researchers
* having a bleeding tendency or a great worry of gastrointestinal bleeding
* with infection requiring antibiotic treatment
* history of immunodeficiency, including HIV positive, organ transplantation and other acquired/congenital immunodeficiency disorders
* patients with Hepatitis B(except inactive carrier) or Hepatitis C
* took part in other clinical studies or is involved in other research projects at present

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2020-08-20 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
nutritional status | From time of randomization to the date of chemotherapy ends or date of death from any cause, whichever came first, assessed up to 6 months
  effect of nutrition-support-team intervention on nutritional status, nutritional risk assessments

SECONDARY OUTCOMES:
chemo-related adverse events | From time of randomization to the date of chemotherapy ends or date of death from any cause, whichever came first, assessed up to 6 months
  amount of chemo-related adverse events
total chemotherapy cycles | From time of randomization to the date of chemotherapy ends or date of death from any cause, whichever came first, assessed up to 6 months
  amount of total cycles of chemotherapy
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 months
  the survival time of patient without progression
adverse events | From time of randomization to one week of the ends of nutritional intervention，assessed up to 7 months
  Amount of adverse events related to nutritional intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiao Zhang, doctor, Study Director — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China